CLINICAL TRIAL: NCT04624399
Title: Phase 2 Study of Neoadjuvant Immune Checkpoint Inhibitors in Urothelial Cancer
Brief Title: Neoadjuvant Immune Checkpoint Inhibitor Treatment in Urothelial Cancer
Acronym: ABACUS-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABACUS-2
Record Dates: First submitted 2020-11-05; First posted 2020-11-10 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Urogenital Cancer
MeSH Terms: conditions — Urogenital Neoplasms | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atezolizumab (Experimental): Patients receive 2 x 3-weekly cycles of Atezolizumab (one infusion on the first day of each cycle) prior to cystectomy surgery.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Patients receive 2 x 3-weekly cycles of Atezolizumab (one infusion on the first day of each cycle) prior to cystectomy surgery.
  Other Names: MPDL3280A

SUMMARY:
This study is being carried out to see if the drug atezolizumab can reduce the size of tumours in patients with types of urothelial cancer before surgery. Atezolizumab is designed to stop a protein called PD-L1 (programmed death-ligand 1) being expressed on the cancer, allowing the immune system to recognise the tumour cells as foreign bodies and attack them. Atezolizumab has been shown to have activity in urothelial cancer which has spread.

There two cohorts for this trial. One cohort will investigate the most common histological type of urothelial cancer (transitional cell carcinoma) outside the bladder, for example in the upper urinary tract. The other cohort will investigate rarer histological subtypes (such as such as squamous cell or adenocarcinoma) of urothelial cancer throughout the entire urinary system.

This study will be recruiting patients from hospitals in the UK, France and Spain. If a patient is eligible for the study and decides to take part, they will receive up to two 3-weekly cycles of atezolizumab. 4-8 weeks after being enrolled, the patient will have an operation to remove the bladder (cystectomy) or the kidney, ureter and part of the bladder (nephroureterectomy or distal ureteral resection) as per normal practice. Following surgery, they will attend three hospital visits (4,12 and 24 weeks after surgery) and their disease progress/survival will be followed over the next 2 years. The clinical team will compare the patient's tumour tissue samples,scan results and blood results from before and after treatment with atezolizumab in order to see how well the drug works and if it is safe. Many of the procedures involved in this study are offered as standard care and participation in this trial will not delay surgery.

ELIGIBILITY:
Inclusion Criteria:

Cohort-Specific Inclusion Criteria • Bladder cohort: Histopathologically confirmed carcinoma of the urothelium (T1 high grade -T4a) in the bladder with mixed or rare histological subtypes such as squamous cell or adenocarcinoma. Patients with mixed histologies are required to have a dominant non- transitional cell pattern.

• UTUC cohort:

Histopathologically confirmed,high grade or high risk upper urinary tract urothelial carcinoma (renal pelvis and ureter). This cohort includes all patients with upper tract malignancy who in the opinion of the investigators qualify for radical surgery (nephroureterectomy or distal ureter resection). Urothelial carcinoma of the upper urinary tract qualifies as high-risk disease if any of the below factors are present:

* Hydronephrosis
* Tumour size >2cm on cross sectional imaging
* High grade cytology
* High grade biopsy
* Multifocal disease
* Variant histology
* Previous radical cystectomy for urothelial cancer of the bladder

All patients undergoing radical surgery with curative intent in the opinion of the investigator are eligible. Radical surgical interventions include nephroureterectomy or distal ureteral resection.

General inclusion criteria:

1. Willing and able to provide written informed consent
2. Ability to comply with the protocol
3. Age ≥ 18 years
4. Residual disease after TURBT or URS (surgical opinion, endoscopy or radiological presence).
5. Fit and planned for radical surgery with curative intent in the opinion of the investigator (according to local guidelines).
6. N0 or M0 disease CT or MRI (within 4 weeks of registration)
7. Representative formalin-fixed paraffin embedded (FFPE) tumour samples with an associated pathology report that are determined to be available and sufficient for central testing.
8. Patients who refuse neoadjuvant cisplatin-based chemotherapy or in whom neoadjuvant cisplatin-based therapy is not appropriate.
9. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
10. Negative pregnancy test within 2 weeks of Day 1 Cycle 1 for female patients of childbearing potential.
11. For female patients of childbearing potential to use a highly effecting form(s) of contraception (i.e. one that results in a low failure rate [<1% per year] when used consistently and correctly) and to continue its use for 90 days after the last dose of atezolizumab.
12. Adequate hematologic and end-organ function within 4 weeks prior to the first study treatment defined by the following:

    1. ANC ≥ 1500 cells/μL (without granulocyte colony-stimulating factor support within 2 weeks prior to Cycle 1, Day 1)
    2. WBC counts > 2500/μL
    3. Lymphocyte count ≥ 500/μL
    4. Platelet count ≥ 100,000/μL (without transfusion within 2 weeks prior to Cycle 1, Day 1)
    5. Haemoglobin ≥ 9.0 g/dL (patients may be transfused or receive erythropoietic treatment to meet this criterion).
    6. AST or ALT,and alkaline phosphatase ≤ 2.5 times the institutional upper limit of normal (ULN) (patients with known Gilbert disease who have serum bilirubin level ≤ 3 × the institutional ULN may be enrolled).
    7. INR and aPTT ≤ 1.5 × the institutional ULN. This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose.
    8. Calculated creatinine clearance ≥ 20 mL/min (Cockcroft-Gault formula)

Exclusion Criteria:

1. Pregnant and lactating female patients.
2. Major surgical procedure within 4 weeks prior to enrolment or anticipation of need for a major surgical procedure during the course of the study other than for diagnosis.
3. Previously intravenous chemotherapy for urothelial cancer.
4. Patients with prior allogeneic stem cell or solid organ transplantation.
5. Prior treatment with CD137 agonists,anti-CTLA-4,anti-programmed death-1 (PD-1),or anti-PD-L1 therapeutic antibody or pathway-targeting agents.
6. Patients must not have had oral or IV steroids for 14 days prior to study entry. The use of inhaled corticosteroids, physiologic replacement doses of glucocorticoids (i.e.,for adrenal insufficiency), and mineralocorticoids (e.g. fludrocortisone) is allowed.
7. Received therapeutic oral or intravenous (IV) antibiotics within 14 days prior to enrolment (Patients receiving prophylactic antibiotics (e.g.,for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible).
8. Administration of a live,attenuated vaccine within 4 weeks prior to enrolment or anticipation that such a live,attenuated vaccine will be required during the study.
9. Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin [IL]-2) within 4 weeks or five half-lives of the drug, whichever is shorter, prior to enrolment.
10. Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 4 weeks prior to enrolment.
11. Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including significant liver disease (such as cirrhosis, uncontrolled major seizure disorder, or superior vena cava syndrome).
12. Malignancies other than UC within 5 years prior to Cycle 1,Day 1,with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, or ductal carcinoma in situ treated surgically with curative intent) or localized prostate cancer treated with curative intent and absence of prostate-specific antigen (PSA) relapse or incidental prostate cancer (Gleason score ≤ 3 + 4 and PSA < 10 ng/mL undergoing active surveillance and treatment naive).
13. Severe infections within 4 weeks prior to enrolment in the study including but not limited to hospitalization for complications of infection, bacteraemia,or severe pneumonia.
14. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within 3 months prior to enrolment, unstable arrhythmias, or unstable angina.
15. History of idiopathic pulmonary fibrosis (including pneumonitis),drug-induced pneumonitis, organizing pneumonia (i.e.,bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan (History of radiation pneumonitis in the radiation field (fibrosis) is permitted).
16. Patients with uncontrolled Type 1 diabetes mellitus. Patients with Type 1 diabetes controlled on a stable insulin regimen are eligible.
17. Patients with active hepatitis infection (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
18. Positive test for HIV
19. Patients with active tuberculosis
20. History of gastrointestinal disorders (medical disorders or extensive surgery) which may interfere with the absorption of the study drug.
21. Uncontrolled hypercalcemia (> 1.5 mmol/L ionized calcium or Ca > 12 mg/dL or corrected serum calcium > the institutional ULN) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab. Patients who are receiving bisphosphonate therapy or denosumab specifically to prevent skeletal events and who do not have a history of clinically significant hypercalcemia are eligible. Patients who are receiving denosumab prior to enrollment must be willing and eligible to receive a bisphosphonate instead while on study.
22. History of autoimmune disease including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.
23. Patients with a history of autoimmune-related hypothyroidism, unless on a stable dose of thyroid-replacement hormone.
24. History of severe allergic, anaphylactic,or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
25. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCRR) | At surgery (4-8 weeks after patient registration)
  No microscopic evidence (pT0/Tis/Cis) of residual disease in the bladder based on histological evaluation of the resected bladder specimen collected during cystectomy (post-treatment) [Bladder Cohort]
  - No microscopic evidence (pT0/Tis/Cis) of residual disease in the renal pelvis or ureter in the resected sample collected during radical surgery for upper tract disease (post-treatment) [UTUC Cohort]
Assessment on immune parameters | Samples acquired at surgery (4-8 weeks after patient registration)
  ynamic changes in T cell subpopulations (CD8 and/or CD3) measured in tumour samples collected pre- and post-treatment.

SECONDARY OUTCOMES:
Evaluate the safety and tolerability of atezolizumab when given in the neoadjuvant setting | Adverse Events will be collated during treatment and up to 24 weeks post-cystectomy or post-radical surgery. Surgical complications will be assessed at the 4wk and 12 week follow-up visits.
  Incidence, nature and severity of Adverse Events graded according to NCI-CTCAE v5.0. Surgical complications will be assessed by the Clavien-Dindo scoring system.
Assess the efficacy of atezolizumab given in the neoadjuvant setting with respect to anti-tumour effects as measured by Investigator assessed radiological response (RR) | Assessed at CT scan pre-surgery.
  RR defined as a ≥30% decrease in tumour diameter from the baseline scan based on local investigator assessments.
Assess the efficacy of atezolizumab given in the neoadjuvant setting with respect to anti-tumour effects based on Investigator assessed disease-free survival (DFS) | Evaluated at 12 weeks, 24 weeks, 12 months, and 24 months post-surgery.
  DFS defined as time between the date of enrolment to first evidence of relapse based on local investigator assessments or death, whichever occurs first.
Assess the efficacy of atezolizumab given in the neoadjuvant setting with respect to overall survival (OS) | Evaluated at 12 weeks, 24 weeks, 12 months, and 24 months post-surgery.
  OS, defined as the time between the date of enrolment and death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Powles, Principal Investigator — Queen Mary University of London
Locations (1):
- Barts and London Hospital NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No